CLINICAL TRIAL: NCT06463743
Title: Metformin as an add-on or Monotherapy in Treatment of Aging People With Multiple Sclerosis (MS): Randomized, Placebo-controlled Pilot Study.
Brief Title: Metformin as an add-on or Monotherapy in Treatment of Aging People With Multiple Sclerosis (MS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Bianca Weinstock-Guttman, Professor of Neurology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00007603; UL1TR001412 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-06-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: metformin
MeSH Terms: conditions — Multiple Sclerosis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- metformin (Experimental): metformin
  Interventions: Drug: metformin
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metformin — metformin
  Arms: metformin
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The goal of the study is to learn about treating older people with multiple sclerosis (MS) with metformin. Metformin may be used as a single therapy or as an add-on therapy. The investigators want to learn:

* The safety and tolerability of metformin extended release (1500 mg/day) as a single therapy or as an add-on therapy in older people with MS compared to placebo
* How well metformin protects the nervous system against injury compared with placebo measured by brain MRI over a 9 month treatment period
* The effect of metformin to protect brain tissue from age and MS related injury when compared to the placebo group over a 9 month treatment period

DETAILED DESCRIPTION:
Specific aims and rationale:

The main aim of this study is to determine the safety of metformin as monotherapy or as an add-on therapy to the disease modifying treatment in aging people with multiple sclerosis (pwMS). While the tolerability of metformin has been studies in the general population, data specific to the MS population is not currently available. Moreover, understanding the gastrointestinal tolerability of metformin when added on MS disease modifying treatment is needed. Secondly, the study aims at understating the potential neuroprotective properties of metformin as measured through magnetic resonance spectroscopy and change in N-acetyl-aspartate (NAA) levels over a 9-month study period. This pilot study will provide valuable insights into the efficacy and safety of add-on or monotherapy metformin therapy as a potential therapeutic approach to address the complex pathophysiology of MS and offer new avenues for promoting neuroprotection along with potential support for neural repair and remyelination in individuals with this debilitating condition. Previous pre-clinical studies have shown that metformin can promote neuroprotection by reducing oxidative stress and inflammation and is able to enhance the reparative mechanisms within the central nervous system (CNS). Currently there are no neuroprotective interventions available for pwMS that directly target the neurodegenerative component of MS, with particular emphasis for the aging MS population. The investigators hypothesize that older pwMS that are treated with metformin will have a significantly lower decline in N-acetylaspartate levels when compared to pwMS not treated with metformin.

ELIGIBILITY:
Inclusion Criteria:

1. age between 55 and 75 years old
2. having a diagnosis of MS based on the latest McDonald criteria
3. non-active disease course (no relapses and no MRI activity) in the last 2 years as determined by the MS provider and based on the 2020 revised clinical course criteria
4. EDSS score <7.0

Exclusion Criteria:

1. inability to undergo MRI scans
2. inability to participate in the study during the study period
3. diabetes or uncontrolled cardiovascular disease
4. unable to consent

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1 year
  The adverse events (AE) will be collected using standardized Adverse Events Form. The severity of the AE will be determined using 5-level grading system where Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of daily living (ADL); Grade 3: Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Life-threatening consequences; urgent intervention indicated; and Grade 5: Death related to AE.
  Additional information regarding the relation to the study medication (related/non related), treatment required (none/drug/non-drug) and the outcome of the AE will be recorded
Percent change in N-Acetyl Aspartate (NAA) in the cortex over 9 months | 9 months
  The MRI scans will be acquired at baseline and 9-month follow-up using magnetic resonance spectroscopy (MRS).

SECONDARY OUTCOMES:
Disability progression as measured with Expanded Disability Status Scale (EDSS) | 1 year
  Disability quantification using Expanded Disability Status Scale (EDSS) (evaluation performed at baseline, 3, 6 and 9 and 12 months). Disability progression will be determined as an increase of 1.0 points in EDSS if the baseline EDSS is <5.5 and increase of 0.5 points in EDSS over the follow-up period if baseline EDSS is ≥5.5 points.
Symbol Digit Modality Test (SDMT) | 1 year
  A neuropsychological assessment will be included using the Brief International Cognitive Assessment in MS (BICAMS) battery at baseline, and 9 months.
  Within the BICAMS battery, the cognitive performance will be evaluated using the Symbol Digit Modalities Test (SDMT)-measuring the correct number match within 90 sec ( higher is better- over 60 normal) . Group difference of 4-points in the SDMT test will be considered as significantly meaningful cognitive difference between the metformin-treated and placebo group.
Brief Visuospatial Memory Test ( BVMT) | 1 year
  correct number of figures out of 6 - immediate and delayed after 20 min
California Verbal Learning Test (CVLT) | 1 year
  Number of words remembered immediate and delayed out of a list of 16 words- (max is 16)
Conventional MRI outcomes | 9 months
  Conventional MRI metrics: lesion burden: number and volume of lesions
Timed 25-foot walk test (T25FWT) | 1 year
  Eval of gait, Change of 20% in the T25FWT (seconds) represents a meaningful change
9-hole peg test (9HPT) | 1 year
  9HPT measured in seconds performed at baseline, 3, 6 and 9 and 12 months. Change of 20% in the 9HPT (seconds) represents a meaningful change
Myelin water fraction (MWF) | 9 months
  Non-conventional MRI metrics : myelin water fraction (MWF)

OTHER OUTCOMES:
Exploratory/tertiary MRI metrics | 9 months
  Exploratory/tertiary MRI metrics assessment of cortical lesion burden using synthetic DIR sequence and perfusion-based imaging using arterial spin labeling (ASL).

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Neurolgy, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No